CLINICAL TRIAL: NCT04842656
Title: Comparison of Active Release Technique and Post Isometric Relaxation in Patients With Piriformis Syndrome
Brief Title: Soft Tissue Techniques in Piriformis Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/00768 Attiq Ur Rehman
Record Dates: First submitted 2021-04-10; First posted 2021-04-13 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-09

CONDITIONS: Piriformis Syndrome
MeSH Terms: conditions — Piriformis Muscle Syndrome

STUDY DESIGN:
Intervention Model Description: Comparison of Active Release Technique and Post Isometric Relaxation in patients with Piriformis Syndrome
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active release technique alongwith conventional treatment (Experimental): Patients in Group A will receive active release technique. ART will be applied with patient in prone lying, knee flexed at 90. The therapist will place his elbow tip on taut band of piriformis and direct pressure is applied, patient is then asked to do internal rotation of hip, in order to achieve lengthening of the muscle. This will be repeated 5-7 times(22).
  Interventions: Other: Active release technique alongwith conventional treatment
- Post isometric relaxation alongwith conventional treatment (Experimental): Patients in group B will receive post isometric relaxation technique. Patient lying in supine position, with the treated leg is placed into flexion at the hip and knee, so that the foot rests on the table lateral to the contra lateral knee (the leg on the side to be treated is crossed over the other). Therapist places one hand on the contra lateral ASIS to prevent pelvic motion, while the other hand is placed against the lateral flexed knee as this is pushed into resisted abduction to contract piriformis (PIR MET). The starting position will be the 1st sign of resistance towards end range. Therapist Force will be same as patient's force. Initial effort is approximately 20% of patient's strength. Duration of contraction is 7-10 seconds with three repetitions(32)
  Interventions: Other: Post isometric relaxation

INTERVENTIONS:
Other: Post isometric relaxation — Patients in group B will receive post isometric relaxation technique. Patient lying in supine position, with the treated leg is placed into flexion at the hip and knee, so that the foot rests on the table lateral to the contra lateral knee (the leg on the side to be treated is crossed over the other). Therapist places one hand on the contra lateral ASIS to prevent pelvic motion, while the other hand is placed against the lateral flexed knee as this is pushed into resisted abduction to contract piriformis (PIR MET). The starting position will be the 1st sign of resistance towards end range. Therapist Force will be same as patient's force. Initial effort is approximately 20% of patient's strength. Duration of contraction is 7-10 seconds with three repetitions
  Arms: Post isometric relaxation alongwith conventional treatment
Other: Active release technique alongwith conventional treatment — Patients in Group A will receive active release technique.ART will be applied with patient in prone lying, knee flexed at 90. The therapist will place his elbow tip on taut band of piriformisand direct pressure isapplied, patient is then asked to do internal rotation of hip, in order to achieve lengthening of the muscle. This will be repeated 5-7 times.
  Arms: Active release technique alongwith conventional treatment

SUMMARY:
The purpose of the study is to compare the effects of active release technique and post isometric relaxation in patients with piriformis syndrome on pain, hip internal rotation range of motion and functional disability. A randomized clinical trial was conducted at Shifa Intl. Hospital, Islamabad. The sample size was 26 calculated through open-epi tool but were recruited 30. The participants were divided into two interventional groups each having 15 participants. The study duration was six months. Sampling technique applied was purposive sampling for recruitment and group randomization using sealed envelope method. Only 35 to 55 years participants with diagnosed piriformis syndrome were included in this study. Tools used in this study are Goniometer, Visual Analogue Scale and lower extremity functional scale. Data was collected at baseline, 3 weeks after sessions and after one month follow up. Data was analyzed through SPSS version 20.

DETAILED DESCRIPTION:
Piriformis syndrome is caused by prolonged or excessive contraction of the piriformis muscle. Because of the close proximity to the sciatic nerve, piriformis syndrome is associated with pain in the buttocks, hips, and lower limbs. Yeoman was the first to describe pain in the sciatic distribution to piriformis syndrome. Many synonyms for the condition are used in the literature, such as ''deep gluteal syndrome'' and ''pelvic outlet syndrome''. It has been suggested that piriformis syndrome is responsible for 5-6% of cases of sciatica. In the majority of cases, piriformis syndrome occurs in middle-aged patients (mean age 38 year). The ratio of female to male patients with piriformis syndrome has been reported as 6:1.

Three specific conditions may contribute to piriformis syndrome:

1. myofascial referred pain from trigger points in the piriformis muscle
2. adjacent muscles, nerve and vascular entrapment by the piriformis muscle at the greater sciatic foramen
3. dysfunction of the sacroiliac joint. Myofascial pain syndrome in the piriformis muscle is well recognized. Gluteal pain is reported to be observed in 97.9% of cases, pain (and paresthesias) in the back, groin, perineum, buttocks, hip, back of the thigh (81.9%),calf (59%),foot, in the rectum (during defecation), and in the area of the coccyx. Low back pain is reported to be observed in 18.1% of cases. Intense pain will occur when the patient sits or squats. Nevertheless, true neurologic findings are not usually present in piriformis syndrome and sensory deficits may be completely absent.

There is no gold standard in diagnosing piriformis syndrome. The physical examination may reveal several of the following well-described signs:

* The piriformis sign, (which presents as tonic external rotation of the affected lower extremity) is reported to be observed in 38.5% of the patients.
* Freiberg's sign involves pain on passive forced internal rotation of the hip in the supine position, thought to result from passive stretching of the piriformis muscle and pressure on the sciatic nerve at the sacrospinous ligament. This test is positive in 56.2% of the patients.
* Pace's sign consists of pain and weakness on resisted abduction and external rotation of the thigh in a sitting position . A positive test is reported to occur in 46.5% of the patient.
* Lasegue's sign involves pain on the affected side on voluntary adduction, flexion, and internal rotation.
* Beatty's maneuver is an active test that involves elevation of the flexed leg on the painful side while the patient lies on the asymptomatic side. Abducting the thigh to raise the knee off the table elicits deep buttock pain in patients with piriformis muscle but back and leg pain in those with lumbar disk disease.
* The Hughes Test (external isometric rotation of the affected lower extremity following maximal internal rotation) may also be positive in piriformis syndrome.
* Gluteal atrophy may be present.Sacroiliac tenderness is reported to be observed in 38.5% of the patients.

Piriformis syndrome causing sciatica usually responds to conservative treatments, including physical therapy, lifestyle modification, pharmacological agents (non-steroidal anti-inflammatory agents, muscle relaxants, and neuropathic pain medication) and psychotherapy. Physiotherapy management for piriformis syndrome includes application of heat therapy and ultrasound therapy in conjunction with stretching of piriformis muscle shows good effect on treatment. Also manual therapy approaches like myofascial release (MFR), muscle energy technique (MET), Active release technique shows beneficial effect on the treatment of soft tissue. The last option is surgical intervention which involves endoscopic decompression of sciatic nerve.

The Active release technique (ART) is a manual therapy used to recover function of soft tissue and in many ways similar to traditional 'Pin and stretch' techniques. Technique works on a variety of muscle, tendon, ligament, fascia and nerve tissues. In this technique deep pressure is applied over the tender point in a shortened position of the muscle and then patient is asked to actively take it in an opposite lengthened position. This will break the adhesions and restores the proper texture, elasticity and functions of soft tissues. There are a variety of studies that imply the value of ART as a treatment method for soft tissue injuries. ART has been used to treat nerve entrapment, tendinopathy, muscle strain, snapping hip syndrome, lateral epicondylitis, impaired range of motion, overuse syndrome, and improve performance and contributed to faster return to activity and decreased treatment time.

Muscle energy technique (MET) is an active muscle based treatment approach that involves the voluntary contraction of a subject's muscle(s) in a precisely controlled direction, against a counterforce provided by the therapist. The MET may be used to decrease pain, stretch tight muscles and fascia, reduce muscle tonus, improve local circulation, strengthen weak musculature and mobilize joint restrictions. The MET is used for achieving tonus release in a muscle before stretching via introduction of an isometric contraction to the affected muscle producing post isometric relaxation. Post isometric relaxation (PIR) is a MET used to relax and lengthen a hypertonic and shortened muscle. This gentle stretching technique is typically used on postural muscles. These muscles often become short and tight and can lead to muscle imbalances. This can limit range of motion and cause joint restrictions.

The effects of ART on gluteus medius for chronic lower back pain and concluded that ART was effective in reducing lower back pain.

ART for ITB syndrome and results showed that ART decreases pain and improves function.

The effects of Neuromuscular therapy and ART on piriformis tightness and concluded that significant improvement was observed in the VAS score and ROM in ART group.

Compared the effectiveness of ART with mulligan bent leg raise for hamstring tightness and concluded that ART was better in improving flexibility and ROM of hamstring.

Compared post isometric relaxation with stretching on piriformis syndrome and concluded that PIR technique group significantly improved in all outcome measures (pain, ROM).

The effects of PIR technique on myofascial tightness of lumbo-pelvic musculature in patients with chronic low back pain and concluded marked improvement in pain and functional disability.

Compared PIR technique with high velocity low amplitude techniques and concluded that both of the techniques are equally effective in managing low back pain.

Compared post isometric relaxation and reciprocal inhibition and concluded that post isometric relaxation is more effective in treating piriformis syndrome than reciprocal inhibition and proposed to follow further in chronic piriformis syndrome.

Currently there is little evidence of relative effects of Active release technique and post isometric relaxation in piriformis syndrome. Both techniques are found to be effective individually in different conditions but no research has been done yet on comparison of active release technique with muscle energy techniques like PIR in piriformis syndrome. Studies of ART on hamstring tightness shows significant immediate effects but the study was on healthy subjects. Effectiveness of ART is evident by one another study but only immediate effects were analyzed. Thus, effective long term follow up is lacking in literature. This present research will fill the gaps by studying the effects of ART and PIR in chronic piriformis syndrome and will help the clinicians with an alternative treatment approach

ELIGIBILITY:
Inclusion Criteria:

* Chronic pain in the buttock and hip area
* Tenderness to palpation over the sciatic notch
* Positive FABER (flexion, abduction, external rotation),FAIR (flexion, adduction, internal rotation) maneuvers.

Exclusion Criteria:

* Malignancies
* History of steroid therapy
* Rheumatoid arthritis/ Osteoarthritis
* Pain medications/ muscle relaxants
* Osteoporosis
* Fracture of femur and hip joint dislocation

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2020-06-30 (Actual); Primary Completion 2021-01-20 (Actual); Study Completion 2021-02-26 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | 6 months
  It is used to measure the intensity or frequency of pain. It ranges on a scale from 0 to 10.
Goniometer | 6 months
  Goniometer is an efficient tool to measure hip range of motion. It measures an angle from 0 to 180.
Lower Extremity Functional Scale | 6 months
  It is a questionnaire containing 20 questions about a persons ability to perform everyday tasks. It minimum score is 0 and maximum score is 80

CONTACTS AND LOCATIONS:
Overall Officials: Lal Gul Khan, MScPT, Principal Investigator — Riphah International University
Locations (1):
- Shifa International Hospital, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Parziale JR, Hudgins TH, Fishman LM. The piriformis syndrome. Am J Orthop (Belle Mead NJ). 1996 Dec;25(12):819-23. PMID 9001677
- [Background] Yeoman W. The Relation Of Arthritis Of The Sacro-Iliac Joint To Sciatica, With An Analysis Of 100 Cases. The Lancet. 1928;212(5492):1119-23.
- [Background] Hopayian K. Sciatica in the community--not always disc herniation. Int J Clin Pract. 1999 Apr-May;53(3):197-8. PMID 10665132
- [Background] Reichel G, Gaerisch F Jr. [Piriformis syndrome. A contribution to the differential diagnosis of lumbago and coccygodynia]. Zentralbl Neurochir. 1988;49(3):178-84. German. PMID 2977249
- [Background] Benson ER, Schutzer SF. Posttraumatic piriformis syndrome: diagnosis and results of operative treatment. J Bone Joint Surg Am. 1999 Jul;81(7):941-9. PMID 10428125
- [Background] Papadopoulos EC, Khan SN. Piriformis syndrome and low back pain: a new classification and review of the literature. Orthop Clin North Am. 2004 Jan;35(1):65-71. doi: 10.1016/S0030-5898(03)00105-6. PMID 15062719
- [Background] Kirkaldy-Willis WH, Hill RJ. A more precise diagnosis for low-back pain. Spine (Phila Pa 1976). 1979 Mar-Apr;4(2):102-9. doi: 10.1097/00007632-197903000-00003. PMID 162546
- [Background] Steiner C, Staubs C, Ganon M, Buhlinger C. Piriformis syndrome: pathogenesis, diagnosis, and treatment. J Am Osteopath Assoc. 1987 Apr;87(4):318-23. No abstract available. PMID 3583849
- [Background] Pace JB. Commonly overlooked pain syndromes responsive to simple therapy. Postgrad Med. 1975 Oct;58(4):107-13. doi: 10.1080/00325481.1975.11714172. No abstract available. PMID 1099564
- [Background] Blaser-Sziede R. Piriformissyndrom-kritische Beurteilung der Literatur und Diskussion der klinischen Zusammenhänge. manuelletherapie. 2006;10(04):159-69
- [Background] Benzon HT, Katz JA, Benzon HA, Iqbal MS. Piriformis syndrome: anatomic considerations, a new injection technique, and a review of the literature. Anesthesiology. 2003 Jun;98(6):1442-8. doi: 10.1097/00000542-200306000-00022. PMID 12766656
- [Background] Hopayian K, Song F, Riera R, Sambandan S. The clinical features of the piriformis syndrome: a systematic review. Eur Spine J. 2010 Dec;19(12):2095-109. doi: 10.1007/s00586-010-1504-9. Epub 2010 Jul 3. PMID 20596735
- [Background] Durrani Z, Winnie AP. Piriformis muscle syndrome: an underdiagnosed cause of sciatica. J Pain Symptom Manage. 1991 Aug;6(6):374-9. doi: 10.1016/0885-3924(91)90029-4. PMID 1880438
- [Background] Freiberg AH. Sciatic pain and its relief by operations on muscle and fascia. Archives of Surgery. 1937;34(2):337-50
- [Background] Fishman SM, Caneris OA, Bandman TB, Audette JF, Borsook D. Injection of the piriformis muscle by fluoroscopic and electromyographic guidance. Reg Anesth Pain Med. 1998 Nov-Dec;23(6):554-9. doi: 10.1016/s1098-7339(98)90080-3. PMID 9840849
- [Background] Kirschner JS, Foye PM, Cole JL. Piriformis syndrome, diagnosis and treatment. Muscle Nerve. 2009 Jul;40(1):10-8. doi: 10.1002/mus.21318. PMID 19466717
- [Background] Hughes SS, Goldstein MN, Hicks DG, Pellegrini VD Jr. Extrapelvic compression of the sciatic nerve. An unusual cause of pain about the hip: report of five cases. J Bone Joint Surg Am. 1992 Dec;74(10):1553-9. No abstract available. PMID 1469018
- [Background] Rodrigue T, Hardy RW. Diagnosis and treatment of piriformis syndrome. Neurosurg Clin N Am. 2001 Apr;12(2):311-9. PMID 11525209
- [Background] Dworkin RH, O'Connor AB, Backonja M, Farrar JT, Finnerup NB, Jensen TS, Kalso EA, Loeser JD, Miaskowski C, Nurmikko TJ, Portenoy RK, Rice ASC, Stacey BR, Treede RD, Turk DC, Wallace MS. Pharmacologic management of neuropathic pain: evidence-based recommendations. Pain. 2007 Dec 5;132(3):237-251. doi: 10.1016/j.pain.2007.08.033. Epub 2007 Oct 24. PMID 17920770
- [Background] Jankovic D, Peng P, van Zundert A. Brief review: piriformis syndrome: etiology, diagnosis, and management. Can J Anaesth. 2013 Oct;60(10):1003-12. doi: 10.1007/s12630-013-0009-5. Epub 2013 Jul 27. PMID 23893704
- [Background] Mujawar JC, Chotai K, Kanase S, Jadhav A. Effectiveness of Neuromuscular Therapy and Active Release Technique in Young Adults with Piriformis Tightness. Indian Journal of Physiotherapy & Occupational Therapy. 2019;13(4):212-7
- [Background] Martin HD, Hatem M, Palmer IJ. Endoscopic sciatic nerve decompression: operative technique. Operative Techniques in Sports Medicine. 2012;20(4):325-32
- [Background] Kage V, Ratnam R. Immediate effect of active release technique versus mulligan bent leg raise in subjects with hamstring tightness: a randomized clinical trial. Int J Physiother Res. 2014;2(1):301-4
- [Background] Moore T. Active release technique for iliotibial band syndrome: A case report: Florida Gulf Coast University; 2014
- [Background] Fryer G, Ruszkowski W. The influence of contraction duration in muscle energy technique applied to the atlanto-axial joint. Journal of osteopathic medicine. 2004;7(2):79-84
- [Background] El Laithy M, Fouda K. Effect of post isometric relaxation technique in the treatment of mechanical neck pain. Physical Therapy and Rehabilitation. 2018;5(1):20
- [Background] Tak S, Lee Y, Choi W, Lee G. The effects of active release technique on the gluteus medius for pain relief in persons with chronic low back pain. Physical Therapy Rehabilitation Science. 2013;2(1):27-30
- [Background] Mahakul B. Effectiveness Of Post Isometric Relaxation Technique And Stretching In Functional Outcome On Piriformis Syndrome: A Randomized Experimental Study 2010
- [Background] Aleksiev A, Kraev T. Postisometric relaxation versus high velocity low amplitude techniques in low back pain. Journal of Orthopaedic Medicine. 2007;29(3):105-8
- [Background] Bose Gnsc, Dusad G. Effect Of Reciprocal Inhibition And Post Isometric Relaxation; Types Of Muscle Energy Technique In Piriformis Syndrome-A Comparative Study
- [Background] Kim JH, Lee HS, Park SW. Effects of the active release technique on pain and range of motion of patients with chronic neck pain. J Phys Ther Sci. 2015 Aug;27(8):2461-4. doi: 10.1589/jpts.27.2461. Epub 2015 Aug 21. PMID 26357426
- [Background] Binkley JM, Stratford PW, Lott SA, Riddle DL. The Lower Extremity Functional Scale (LEFS): scale development, measurement properties, and clinical application. North American Orthopaedic Rehabilitation Research Network. Phys Ther. 1999 Apr;79(4):371-83. PMID 10201543